CLINICAL TRIAL: NCT04092985
Title: Feasibility and Reliability of Smart Watch iECG for the Detection of Cardiac Arrhythmias (The Leipzig Apple Heart Rhythm Study)
Brief Title: Smart Watch iECG for the Detection of Cardiac Arrhythmias
Status: Completed | Type: Observational
Sponsor: Helios Health Institute GmbH (Other)
Collaborators: Heart Center Leipzig - University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-0157
Record Dates: First submitted 2019-09-16; First posted 2019-09-17 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Arrhythmias, Cardiac; Atrial Fibrillation
Keywords: Arrhythmias, Cardiac; Cardiovascular App; Rhythm monitoring
MeSH Terms: conditions — Arrhythmias, Cardiac; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Patients suspected with Cardiac Arrhythmia: iECG + 12-lead ECG recording in patients suspected with any type of cardiac arrhythmias at the time of recruitment
  Interventions: Device: iECG recording

INTERVENTIONS:
Device: iECG recording — iECG tracings will be recorded simultaneously, starting and ending at the same time as the standard 12-lead ECG, using the built-in sensors of a smart watch (Apple Watch Series 4) with the ECG application

SUMMARY:
This study aims to assess the feasibility and reliability of smart watch iECG provided by the Apple Watch/Apple iPhone for the detection of different cardiac arrhythmias. In this study, results from a 12-lead ECG will be set as the gold standard for the arrhythmia diagnosis, and results from the smart watch iECG (Apple watch/Apple iPhone application and Cardiologist's interpretations) as the index tests. The iECG tracings will be recorded simultaneously, starting and ending at the same time as the standard 12-lead ECG, using the built-in sensors of a smart watch (Apple Watch Series 4) with the ECG application.

DETAILED DESCRIPTION:
This diagnostic accuracy study is an investigator-initiated trial to evaluate the value of a smart watch-based iECG for detection of cardiac arrhythmias.

iECG tracings will be recorded simultaneously, starting and ending at the same time as the standard 12-lead ECG, using the built-in sensors of a smart watch (Apple Watch Series 4) with the market version of the ECG application (Apple Inc., California). Participants will be advised to lie down in a supine position and breathe spontaneously. All recording will be done by trained study personnel.

All iECG and 12-lead ECG recordings will be presented in PDF format as our references. Saved formats will be transferred to our Telemonitoring Center for further analysis and processing.

Results from a 12-lead ECG will be considered as the gold standard for the measurement of heart rhythms and the arrhythmia diagnosis. All 12-lead ECGs recordings will be analyzed by 2 blinded cardiologists and will be categorized as "Sinus rhythm", "High or low heart rate", "Atrial fibrillation", or "Inconclusive". Besides, cardiologists will report ECG wave's characteristics as well as any other possible diagnosis including "Superior ventricular tachycardia", "Ventricular tachycardia", "Atrial flutter", and "other types: other possible arrhythmias". In the case of uncertainties, a third cardiologist will be consulted, blinded for initial diagnoses.

The iECG recordings (test index) will be interpreted and reported in two different ways:

1. By using HealthKit Framework (Apple Watch and Apple iPhone applications): After a successful iECG recording with the Apple watch, iECGs will be transmitted by the ECG application to the iPhone. The Health App (Apple Inc., California) will receive, process and store the iECGs on the iPhone and will present one of the following results on the iPhone screen automatically: "Sinus rhythm", "High or low heart rate", "Atrial fibrillation", or "Inconclusive". Besides, the mean heart rate will be recorded, which will be automatically calculated by the Health App.
2. By cardiologist: All iECGs will be analyzed by 2 blinded cardiologists. They will report their findings in the following categorize: "Sinus rhythm", "High or low heart rate", "Atrial fibrillation", or "Inconclusive". Besides, they will report ECG wave's characteristics as well as any other possible diagnosis including "Superior ventricular tachycardia", "Ventricular tachycardia", "Atrial flutter", and "other types: other possible arrhythmias". In the case of uncertainties, a third cardiologist will be consulted, blinded for initial diagnoses.

ECG wave's characteristics: The following variables will be measured as the iECG and 12-lead ECG waves' characteristics. Three randomly chosen heartbeats will be considered to measure each wave or interval, and the mean of these 3 measurements will be used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged≥22 years at the time of eligibility screening will be included.
* Patients with known cardiac arrhythmias; i.e. AF before and after cardioversion, hemodynamically stable Bradycardias, SVT and VT during EP procedures and implants can also be included

Exclusion Criteria:

- Pregnancy

Min Age: 22 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All individuals who had been admitted to the Department of Electrophysiology, Leipzig Heart Center
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Level of agreement between the cardiologist's interpretations of the 12-lead ECG and the ECG App interpretation results | Baseline
Level of agreement between the cardiologist's interpretations of the 12-lead ECG and iECG | Baseline
Level of agreement between the cardiologist's interpretations of the iECG and the ECG App interpretation results | Baseline

SECONDARY OUTCOMES:
Proportion of participants that remain in arrhythmia diagnosis, from the positive diagnosis from the iECG to the performed 12-lead ECG | Baseline
Proportion of interpretable and non-interpretable iECGs | Baseline
Sensitivity and specificity of screening tests for cardiac arrhythmias identification using: cardiologists interpretation of iECG (index test) and 12-lead ECGs (reference test) | Baseline
Sensitivity and specificity of screening tests for cardiac arrhythmias identification using: ECG App interpretation results (index test) and 12-lead ECGs (reference test) | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Bollmann, MD, PhD, Study Chair — Heart Center Leipzig at University of Leipzig, Leipzig Heart Institute, Germany
Locations (1):
- Andreas Bollmann, Leipzig, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Behzadi A, Sepehri Shamloo A, Mouratis K, Hindricks G, Arya A, Bollmann A. Feasibility and Reliability of SmartWatch to Obtain 3-Lead Electrocardiogram Recordings. Sensors (Basel). 2020 Sep 7;20(18):5074. doi: 10.3390/s20185074. PMID 32906661